CLINICAL TRIAL: NCT03348072
Title: Comparative Study of Survival and Long-term Quality of Life After Cardiac Surgery in Patients Who Are Jehovah's Witnesses
Status: Completed | Type: Observational
Sponsor: Pierre Wauthy (Other)
Responsible Party: Sponsor-Investigator, Pierre Wauthy, Head of clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-QoL Jehovah
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Cardiac Surgery
MeSH Terms: interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Jehovah's witnesses: Jehovah's witnesses having undergone cardiac surgery between 1991 till 2012. Blood perfusions refused.
  Interventions: Procedure: Cardiac surgery
- Control: Paired control group, twice as big as the experimental group. Pairing criteria: age, sex, type of surgery performed. The control group must accept blood transfusions.
  Interventions: Procedure: Cardiac surgery

INTERVENTIONS:
Procedure: Cardiac surgery — Cardiac surgery

SUMMARY:
This is a comparative study on the survival and long-term quality of life of Jehovah's witnesses having undergone a cardiac surgery and having refused blood transfusions for religious reasons. This group will be compared with two other groups having no restrictions on this subject.

The purpose of the study is to evaluate the impact of this decision on survival and postoperative quality of life, in the long term.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery with extra corporeal blood circulation
* Informed consent given

Exclusion Criteria:

* Dementia (must be able to answer the questionnaire)
* Control group: refusal of blood transfusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Jehovah's withnesses having undergone cardiac surgery between 1991 till 2012 (blood perfusions refused) and paired control group having had the same surgical interventions (blood perfusions allowed)
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Quality of life (score) | Evaluated once by means of a phone contact performed in 2016, irrespective of the date the surgery was performed
  Score computed with the "MacNew Heart Disease health-related quality of life instrument".The MacNew is a valuable tool for assessing and evaluating health related quality of life in heart disease patients. It consists of 27 questions, falling into 3 possible domains: physicial limitation capacity (13 questions), emotional domain (14 questions), social domain (13 questions), symptom related (5 questions). The time frame for the MacNew is the previous two weeks. Scoring of the MacNew is simple: one score in each domain and a global score (4 scores). The maximum possible score in any domain is 7 [high HRQL] and the minimum is 1 [poor HRQL].The global score is calculated as the average over all scored items unless one of the domains is completely missing.
Survival rate | Evaluated once by means of a phone contact performed in 2016, irrespective of the date the surgery was performed
  Survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Wauthy, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wauthy P, Pierrakos C, Chebli L, Tortora R. Long-term survival and quality of life in Jehovah's witnesses after cardiac surgery: a case control study. BMC Cardiovasc Disord. 2019 Mar 29;19(1):73. doi: 10.1186/s12872-019-1061-z. PMID 30922241